CLINICAL TRIAL: NCT01277939
Title: Computerized Psychosocial Treatment for Offenders With Substance Use Disorders
Brief Title: CPT for Offenders With SUD
Acronym: CPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Development and Research Institutes, Inc. (Other)
Collaborators: University of California, Los Angeles (Other); Temple University (Other); University of Kentucky (Other); University of Miami (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NDRI-612; 1RC2DA028967 (NIH)
Record Dates: First submitted 2011-01-12; First posted 2011-01-17 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Computer-assisted, Evidence-based Psychosocial Intervention; for Substance Abuse Treatment
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Therapeutic Education System (TES) (Experimental): Experimental (E) condition, the Therapeutic Education System (TES) delivered via effective informational technologies and multimedia learning tools.
  Interventions: Behavioral: Therapeutic Education System (TES)
- Standard Care (Active Comparator): The Control (C) condition, Standard Care, consisting of psycho-educational and psycho-social approaches to substance use disorders (commonly offered in prison settings) delivered by counselors in group formats.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Therapeutic Education System (TES) — Therapeutic Education System (TES) is an interactive, computer-based, psychosocial treatment program. TES is theoretically grounded in evidence-based psychosocial treatments (Community Reinforcement Approach and Cognitive Behavioral Therapy).
  Arms: Therapeutic Education System (TES)
Behavioral: Standard Care — Psycho-educational and psycho-social approaches to substance use disorders (commonly offered in prison settings) delivered by counselors in group formats.
  Arms: Standard Care

SUMMARY:
This study will evaluate the comparative effectiveness of Therapeutic Education System (TES), a computer-based, psychosocial treatment program, relative to standard care when offered to individuals with substance use disorders in prison settings. The study will assess the comparative effectiveness of these interventions primarily by examining changes in: (1) substance use (e.g., weeks of abstinence), (2) HIV risk behavior (evaluated as both sex-related and drug-related HIV risk behavior) and (3) reincarceration rates. The study will also examine the extent to which these interventions improve psychosocial functioning (e.g., employment, health, and psychological status) and quality of life, and promote relevant skills acquisition (e.g., improve communication skills, reduce "criminal thinking"). The investigators predict significantly better outcomes for E vs. C due to TES' research-based content and use of proven informational technologies.

DETAILED DESCRIPTION:
The majority of individuals in criminal justice settings across the U.S. have a critical need for science-based, psychosocial treatment that targets substance use and HIV risk behavior. The investigative team has developed and demonstrated the efficacy of an interactive, computer-based, psychosocial treatment pro-gram, the Therapeutic Education System (TES), which can answer this need. TES is theoretically grounded in evidence-based psychosocial treatments (Community Reinforcement Approach and Cognitive Behavioral Therapy), and employs state-of-the-art, proven informational technologies and multimedia learning tools to promote skills acquisition, experiential learning and behavioral change. This computer-based therapeutic tool allows complex interventions to be delivered with fidelity to the evidence-based model and at low cost due to its self-directed nature (e.g., minimal staff time/training needed), thus offering considerable potential for future sustainability and dissemination within criminal justice systems.

The study employs random assignment of incarcerated male and female offenders with substance use disorders (N=526) to either (1) TES (N=263), or (2) Standard Care (N=263), in a multi-site trial conducted in 8 prison substance abuse programs. Along with NDRI (the applicant organization), the collaborating study sites (University of California Los Angeles, Temple University, and the University of Kentucky) operate Research Centers that belong to the Criminal Justice Drug Abuse Treatment Studies (CJDATS) network, a NIDA-funded cooperative agreement, which has established relationships with criminal justice partners from Departments of Corrections across the U.S. Aim 1 is to test the comparative effectiveness of TES vs. Standard Care on measures of drug use (e.g., weeks of abstinence) and HIV risk behavior (both sex-related and drug-related HIV risk behavior) at 3- and 6-months post prison discharge, as well as on reincarceration rates using official Department of Corrections records. Aim 2 is to evaluate the cost and cost-effectiveness of TES relative to standard care. The investigators predict that TES will be significantly more effective and cost effective than Standard Care.

The project is significant in its use of an innovative, computer-based technology and in its potential to produce a major increase in the effective and cost-effective delivery of science-based psychosocial treatment to substance-abusing offenders in prison, and thereby make a considerable public health contribution. Thus, funding the proposed 2-year project can markedly accelerate the pace and achievement of research and dissemination efforts to meet the needs of the U.S. correctional community by providing effective and practical treatment interventions for its large substance-abusing population.

ELIGIBILITY:
Inclusion Criteria:

* individual's parole eligibility date or mandatory release date must be scheduled to occur within a minimum of 4 months (to allow intake an treatment to be completed) and a maximum of 6 months (to ensure that their release follows completion of their treatment such that sufficient time remains for post-prison follow-up interviews to occur within the two-year project timeframe)
* the state criminal justice system must have identified the individual to have a substance use disorder that requires a substance abuse intervention
* the individual must give their informed consent

Exclusion Criteria:

* the individual must not already be participating in substance abuse treatment
* the individual must speak English, as TES is now only available in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Time Line Follow Back for Drug and Alcohol Use (Sobell et al., 1996) | 6 months post-prison release
  Measure for substance use.
Urinalysis | 6 months post-prison release
  To detect any change in illicit drug use.
Risk Behavior Survey (Booth et al., 1993) | 6 months post-prison release
  To assess both drug-related and sex-related HIV risk behavior.
DOC record systems | At an average of 11 months post-prison release
  To provide the reincarceration status of each participant.

SECONDARY OUTCOMES:
Coping Strategies Scale | 6 months post-prison release
  Measures skills acquisition, such as problem solving and dealing with urges to use substances of abuse (Litt et al., 2005), and psychosocial functioning
Addiction Severity Index-Lite | 6 months post-prison release
  Measures areas of health status improvement, psychological status, family/social relationships, and employment. (www.tresearch.org)
The Treatment Services Review instrument (McLellan et al., www.tresearch.org) | 6 months post-prison release
  Used to investigate the role of treatment services received post-release (in aftercare).
Brief Drug Abuse Treatment Cost Analysis Program (BriefDATCAP) | 6 months post-prison release
  Measures for the cost effectiveness analyses.
EuroQol EQ5D (QOL) (the EuroQol Group, 1990) | 6 months post-prison release
  Describes and value health-related quality of life and for constructing Quality-Adjusted Life Year estimates (QALYs).

CONTACTS AND LOCATIONS:
Overall Officials: Stan Sacks, PhD, Principal Investigator — National Development & Research Institutes
Locations (10):
- United States (10):
  - Colorado Territorial Correctional Facility, Cañon City, Colorado
  - Four Mile Correctional Center, Cañon City, Colorado
  - Fremont Correctional Facility, Cañon City, Colorado
  - Denver Women's Correctional Facility, Denver, Colorado
  - Trinidad Correctional Facility, Model, Colorado
  - La Vista Correctional Facility, Pueblo, Colorado
  - Sterling Correctional Facility, Sterling, Colorado
  - Blackburn Correctional Complex, Lexington, Kentucky
  - SCI Cambridge Springs, Cambridge Springs, Pennsylvania
  - Airway Heights Corrections Center, Airway Heights, Washington